CLINICAL TRIAL: NCT06371170
Title: Rivaroxaban for Intracardiac Thrombosis in the Pediatric Population at Different Cardiac Sites
Brief Title: Rivaroxaban for Intracardiac Thrombosis in the Pediatric Population
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Responsible Party: Principal Investigator, Francesco Bianco, Principal Investigator, Azienda Ospedaliero, Universitaria Ospedali Riuniti
Other Study IDs: CCPC- 001/22
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Intracardiac Thrombus
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rivaroxaban — Oral anticoagulation
  Other Names: Xarelto

SUMMARY:
The goal of this observational study is to determine the efficacy of rivaroxaban treatment for intracardiac thrombi resolution in pediatric patients (< 16 years old) diagnosed with intracardiac thrombosis. The main question it aims to answer is: Does rivaroxaban treatment resolve the thrombosis during a 3-month treatment?

Participants already taking rivaroxaban as part of their regular medical care for thrombosis resolution. They will undergo monthly visits to check that the treatment is progressing correctly and that no major bleeding has occurred. After 3 months of treatment, they will repeat the radiological imaging investigation to verify the actual resolution of the thrombosis.

DETAILED DESCRIPTION:
The Investigators will enroll all the consecutive pediatric patients (< 16 years old) treated with rivaroxaban (dosage based on patient's body weight - 0.9 mg/Kg/Day) due to intracardiac thrombosis (ICT) suspected by echocardiography and confirmed with cardiac computed tomography (CCT) or magnetic resonance (CMR) imaging. All the participants will be treated with enoxaparin for 7 days before the rivaroxaban implementation. The treatment will last for 3 months.

The participants will undergo monthly visits to check that the treatment is progressing correctly and that no major bleeding has occurred. Bleeding severity will be assessed utilizing the Bleeding Assessment Scale in Critically Ill Children (BASIC). CCT/CMR will be repeated to confirm the thrombosis resolution. After 3 months of treatment, they will repeat the radiological imaging investigation to verify the effective resolution of the thrombosis, or it will be continued for another 3 months if there is no resolution of the thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Intracardiac thrombosis demonstration at echocardiography and CMR/CCT confirmation
* Given informed consent from the parents or tutors

Exclusion Criteria:

* < 38 weeks of gestational birth
* < 10 days of oral feeding and body weight
* < 2.6 Kg
* Any major or clinically relevant bleeding event or abnormal coagulation test results within 10 days prior to the enrollment for the whole population

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients (neonates and pediatrics) diagnosed with intracardiac thrombosis at any possible cardiac site (right/left ventricle, right/left atria, or auricola).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Thrombus resolution | 3 months
  Rate of intracardiac thrombus resolution at CMR/CCT imaging

SECONDARY OUTCOMES:
Bleeding | 3 months
  Rate of major bleeding utilizing the BASIC bleeding score

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bianco, M.D., Ph.D., Principal Investigator — AOU - Ospedali Riuniti Ancona
Locations (1):
- CCPC, Ancona, The Marches, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Upon request, the data will be shared depending on the requests

REFERENCES:
- [Background] Ozkutlu S, Ozbarlas N, Ozme S, Saraclar M, Gogus S, Demircin M. Intracardiac thrombosis diagnosed by echocardiography in childhood: predisposing and etiological factors. Int J Cardiol. 1993 Jul 15;40(3):251-6. doi: 10.1016/0167-5273(93)90008-5. PMID 8225659
- [Background] Yang JY, Williams S, Brandao LR, Chan AK. Neonatal and childhood right atrial thrombosis: recognition and a risk-stratified treatment approach. Blood Coagul Fibrinolysis. 2010 Jun;21(4):301-7. doi: 10.1097/MBC.0b013e3283333c7c. PMID 20305543
- [Background] Nellis ME, Tucci M, Lacroix J, Spinella PC, Haque KD, Stock A, Steiner ME, Faustino EVS, Zantek ND, Davis PJ, Stanworth SJ, Cholette JM, Parker RI, Demaret P, Kneyber MCJ, Russell RT, Stricker PA, Vogel AM, Willems A, Josephson CD, Luban NLC, Loftis LL, Leteurtre S, Stocker CF, Goobie SM, Karam O; Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network; and the Pediatric Critical Care Blood Research Network (BloodNet). Bleeding Assessment Scale in Critically Ill Children (BASIC): Physician-Driven Diagnostic Criteria for Bleeding Severity. Crit Care Med. 2019 Dec;47(12):1766-1772. doi: 10.1097/CCM.0000000000004025. PMID 31567407
- [Background] Male C, Lensing AWA, Palumbo JS, Kumar R, Nurmeev I, Hege K, Bonnet D, Connor P, Hooimeijer HL, Torres M, Chan AKC, Kenet G, Holzhauer S, Santamaria A, Amedro P, Chalmers E, Simioni P, Bhat RV, Yee DL, Lvova O, Beyer-Westendorf J, Biss TT, Martinelli I, Saracco P, Peters M, Kallay K, Gauger CA, Massicotte MP, Young G, Pap AF, Majumder M, Smith WT, Heubach JF, Berkowitz SD, Thelen K, Kubitza D, Crowther M, Prins MH, Monagle P; EINSTEIN-Jr Phase 3 Investigators. Rivaroxaban compared with standard anticoagulants for the treatment of acute venous thromboembolism in children: a randomised, controlled, phase 3 trial. Lancet Haematol. 2020 Jan;7(1):e18-e27. doi: 10.1016/S2352-3026(19)30219-4. Epub 2019 Nov 5. PMID 31699660
- [Background] Agarwal S, Abdelghani E, Stanek JR, Sankar A, Cua CL, Kerlin BA, Rodriguez V. Intracardiac thrombi in pediatrics: anticoagulation approach and treatment outcomes. Res Pract Thromb Haemost. 2023 Nov 24;7(8):102266. doi: 10.1016/j.rpth.2023.102266. eCollection 2023 Nov. PMID 38193068
- [Derived] Cappelletti D, Bianco F, Bucciarelli V, Raffaelli E, Bordignon L, Di Cesare G, Bucciarelli B, Bacchiocchi A, Manini C, Merlino E, Filippelli S, Lionetti ME. Comparison of rivaroxaban with warfarin for intracardiac thrombosis in the pediatric population at different cardiac sites: Early experience of anticoagulation approach and treatment outcomes. Thromb Res. 2025 Sep;253:109397. doi: 10.1016/j.thromres.2025.109397. Epub 2025 Jul 5. PMID 40628107